CLINICAL TRIAL: NCT04156113
Title: The Effect of an Acute Maximal Exercise on Serum Uncoupling Protein-1 Level and the Role of Uncoupling Protein-1-3826 A/G Polymorphism
Brief Title: Effect of an Exercise on Serum Uncoupling Protein-1 Level and the Role of Uncoupling Protein-1-3826 A/G Polymorphism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Jeffry Roy Chauchat, Senior instructor, Eastern Mediterranean University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-10.2/56
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Uncoupling Protein-1; Polymorphism, Restriction Fragment Length; Irisin
Keywords: Beige fat cell; Fat tissue; Athletes; Sedentary people; Irisin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Athletes Group (Experimental): The athletes group will be composed of healthy, non obese (body mass index < 30), male basketball, volleyball and handball players aged between 18 and 35 years who have been training regularly for at least 3 months. Participants must not be regular consumer of cigarettes, alcohol, drugs and antioxidant substances.
  Intervention: Yo-Yo intermittent recovery test (level 1) is administered.
  Interventions: Other: Yo-Yo intermittent recovery test (level 1)
- Sedentary Group (Experimental): The sedentary group will be composed of healthy, non obese (body mass index < 30), male aged between 18 and 35 years who have not been training regularly for at least 3 months. Participants must not be regular consumer of cigarettes, alcohol, drugs and antioxidant substances.
  Intervention: Yo-Yo intermittent recovery test (level 1) is administered.
  Interventions: Other: Yo-Yo intermittent recovery test (level 1)

INTERVENTIONS:
Other: Yo-Yo intermittent recovery test (level 1) — The Yo-Yo intermittent recovery test (level 1) will be administered once.

SUMMARY:
This study aims to determine the effect of an acute maximal exercise on serum uncoupling protein-1, irisin, interleukin 6 levels, and on blood lipid and lipoprotein concentrations. This study also evaluates the role of uncoupling protein-1-3826 A/G polymorphism on this eventual effect.

Therefore, this study hypothesizes that:

H01: Sedentary people and athletes' serum uncoupling protein 1, irisin, and interleukine 6 levels are different before and after an acute maximal exercise.

H02: Sedentary people and athletes' basal serum uncoupling protein 1 levels are associated with uncoupling protein 1-3826 A/G polymorphism.

H03: Uncoupling protein 1-3826 A/G polymorphism has a modifying role in the effect of maximal exercise on serum uncoupling protein 1 levels.

H04: Sedentary people and athletes' basal serum lipid and lipoprotein levels are associated with uncoupling protein 1-3826 A/G polymorphism.

H05: Uncoupling protein 1-3826 A / G polymorphism has a modifying role in the effect of maximal exercise on serum lipid and lipoprotein levels.

ELIGIBILITY:
Inclusion Criteria:

* Athletes group:

  * Must be basketball, or volleyball, or handball players.
  * Must be subjects who have been training regularly for at least 3 months.
* Sedentary group:

  * Must be subjects who have not been training regularly for at least 3 months.
* For both groups:

  * Healthy.
  * Non obese (body mass index < 30).
  * Aged between 18 and 35 years.

Exclusion Criteria:

* For both groups:

  * Being regular consumer of cigarettes, alcohol, drugs and antioxidant substances.
  * Being obese (body mass index > 30).
  * Having an acute or chronic injury which is limiting physical performance.
  * Having a disease (anemia, infection...) detected from the biochemical analysis of the blood samples.
  * Being injured or sick during the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Change from the baseline serum uncoupling protein 1 level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples were taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Uncoupling protein 1 analyzes were performed in the laboratory.
Change from the baseline serum irisin level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Irisin analyzes were performed in the laboratory.
Uncoupling protein-1-3826 A/G polymorphism determination | 15 minutes before the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples were taken 15 minutes before the Yo-Yo intermittent recovery test (level 1). Polymorphism was determined in the laboratory.

SECONDARY OUTCOMES:
Change from the baseline serum interleukin-6 level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Interleukine-6 analyzes were performed in the laboratory.
Change from the baseline serum nitric oxide level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Nitric oxide analyzes were performed in the laboratory.

OTHER OUTCOMES:
Change from the baseline serum C reactive protein level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. C reactive protein analyzes were performed in the laboratory.
Change from the baseline serum creatine kinase level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Creatine kinase analyzes were performed in the laboratory.
Change from the baseline serum alanine aminotransferase level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Alanine aminotransferase analyzes were performed in the laboratory.
Change from the baseline serum aspartate aminotransferase level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Aspartate aminotransferase analyzes were performed from serum samples in the Medical Biochemistry Laboratory of the Ege University Faculty of Medicine.
Change from the baseline hemogram test at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Hemogram test analyzes were performed in the laboratory.
Change from the baseline at serum glucose level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Glucose analyzes were performed in the laboratory.
Change from the baseline serum urea level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Urea analyzes were performed in the laboratory.
Change from the baseline serum creatinine level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Creatinine analyzes were performed in the laboratory.
Change from the baseline serum total cholesterol level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Total cholesterol analyzes were performed in the laboratory.
Change from the baseline serum low density lipoprotein level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Low density lipoprotein analyzes were performed in the laboratory.
Change from the baseline serum high density lipoprotein level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. High density lipoprotein analyzes were performed in the laboratory.
Change from the baseline serum triglyceride level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Triglyceride analyzes were performed in the laboratory.
Change from the baseline serum total antioxidant level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Total antioxidant analyzes were performed in the laboratory.
Change from the baseline serum total oxidant level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Total oxidant analyzes were performed in the laboratory.
Change from the baseline heparin plasma thiobarbituric acid reactive substances level at 3 minutes post Yo-Yo intermittent recovery test (level 1) | 15 minutes before and 3 minutes after the Yo-Yo intermittent recovery test (level 1)
  Volunteers' postprandial venous blood samples was taken 15 minutes before the Yo-Yo intermittent recovery test (level 1) and 3 minutes post test. Thiobarbituric acid reactive substances analyzes were performed in the laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Turgay, Assoc. Prof, Study Chair — Ege University, Faculty of Sports Science
Locations (1):
- Ege University Faculty of Sport Sciences, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided